CLINICAL TRIAL: NCT04152460
Title: Clinical Assessment of Thermo-Viscous Conventional Bulk-fill Resin Composite in Proximal Compound Posterior Restorations : A Randomized Controlled Clinical Trial
Brief Title: Clinical Assessment of Preheated Versus Conventional Bulk Fill Resin Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Atef Ahmed Ibrahim, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD-CU-2019-10-29
Record Dates: First submitted 2019-11-03; First posted 2019-11-05 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Clinical Significance of Thermo-Viscous Composite
Keywords: Bulk-fill resin Composite; Thermo-Viscous resin Composite; Proximal Compound Cavities

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermo-Viscous preheated bulk fill resin composite (Active Comparator): Viscalor Despenser (Preheating dispenser for composite Viscalor Bulk Caps)
  Interventions: Device: Viscalor Bulk (VOCO,Cuxhaven)
- Conventional Bulk Fill resin Composite (Placebo Comparator): GrandioSo X-tra (Voco,Cuxhaven
  Interventions: Other: Grandioso x-tra

INTERVENTIONS:
Device: Viscalor Bulk (VOCO,Cuxhaven) — Viscalor Despenser (Preheating dispenser for composite Viscalor Bulk Caps)
  Arms: Thermo-Viscous preheated bulk fill resin composite
Other: Grandioso x-tra — Nanohybrid Bulk Resin Composite
  Arms: Conventional Bulk Fill resin Composite

SUMMARY:
A Randomized clinical trial to evaluate the clinical assessment of thermo-viscous versus conventional bulk fill resin composite in proximal compound posterior teeth.The null hypothesis is that there is no difference between thermo-viscous and conventional bulk fill resin composite.

DETAILED DESCRIPTION:
Despite the improvements in resin composite materials some drawbacks still compromise the longevity of resin composite the most frequent reported limitations are related to polymerization shrinkage , to overcome these problem attempts have been made to improve the mechanical properties , the high viscosity and material stickiness as well as adaptation of the material to the walls was difficult and unpredictable .

Preheating is a method that decreases resin composite viscosity results in better adaptation and wettability of the prepared cavity walls reducing the microleakage.

A new approach based on therm-viscous technology Viscalor bulk (VOCO, Cuxhaven ) a high Viscous composite material at room and body temperature by heating to 68 C converted to flowable consistency.

Preheating composite regarding the lab research have significant clinical advantages as better adaptation reduced leakage and increase of mechanical properties .

Follow up Period will be 1 year , Evaluation will be done at baseline , after 6 months and 12 months .

ELIGIBILITY:
Inclusion Criteria:

* Patients aging more than 18 years .
* Patients with a high level of oral hygiene.
* Patients having at least 12 posterior teeth in occlusion.
* Patients with good likelihood of recall availability.

Tooth Inclusion :

* Permanent premolars and molars.
* Moderate to deep compound class II cavities.
* well formed fully erupted .
* Vital with positive reaction to cold and hot stimulus.

Exclusion Criteria:

* Participants with general systematic illness.
* Pregnant or lactating females.
* Concomitant participation in another research study.
* Inability to comply with study procedures.
* Heavy Bruxism habits.
* Patients receiving Orthodontic treatment.
* last experience with allergic reactions against any component of used materials .

Tooth exclusion :

* Non vital teeth.
* Secondary carious lesions.
* Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Integrity | 1 year
  Modified US Public Health Service Criteria (USPHS)

SECONDARY OUTCOMES:
Clinical Evaluation of restoration ( Marginal discoloration,secondary caries and Postoperative Sensitivity ) | 1 year
  Modified US Public Health Service Criteria (USPHS)

CONTACTS AND LOCATIONS:
Overall Officials: Olfat Hasanen, Principal Investigator — Cairo University
Locations (1):
- Yasmin, Cairo, Mokattam, Egypt

IPD SHARING:
Plan to Share IPD: No